CLINICAL TRIAL: NCT03697356
Title: A Multicenter Prospective Phase II Study of Rituximab Combined, Lenalidomide, Dexamethasone Followed by Lenalidomide Maintenance in Patients With Newly Diagnosed Waldenström's Macroglobulinemia
Brief Title: R-VRD Followed by Lenalidomide Maintenance in Patients With Waldenstrom's Macroglobulinemia
Acronym: Ballondor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kosin University Gospel Hospital (Other)
Responsible Party: Principal Investigator, Ho Sup Lee, MD, PhD. associate professor., Kosin University Gospel Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ballondor
Record Dates: First submitted 2018-10-01; First posted 2018-10-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Waldenström's Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Lenalidomide; Bortezomib; Rituximab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rituximab&Bortezomib&Lenalidomide&Dexamethasone (Experimental): Rituximab&Bortezomib&Lenalidomide&Dexamethasone
  Interventions: Drug: Lenalidomide, Bortezomib, Rituximab, Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide, Bortezomib, Rituximab, Dexamethasone — step 1; R-VRD induction : rituximab, bortezomib, lenalidomide, and dexamethasone induction
  * Rituximab 375 mg/m2 intravenous on day 1
  * Bortezomib 1.3mg/m2 subcutaneous on day 1, 8, 15
  * Lenalidomide 15mg p.o on day 1-21
  * Dexamethasone 20 mg/m2 intravenous or p.o on day 1-4
  Step 2 ; Maintenance Beginning 8 weeks after completion of induction therapy, patients receive lenalidomide 10mg once day 1-21 for 4 weeks. Treatment repeats every 1 months for 24 months.

SUMMARY:
A multicenter prospective phase II study of rituximab combined, lenalidomide, dexamethasone followed by lenalidomide maintenance in patients with newly diagnosed Waldenström's macroglobulinemia (Ballondor trial)

DETAILED DESCRIPTION:
Most patients with Waldenstrom's Macroglobulinemia are rare, and most studies are based on Phase II clinical studies, so the most effective regimen has not been established. However, in patients without experience of treatment with rituximab monotherapy targeting CD20 antigen expressed on lymphocytic cells, the response rate is reported to be approximately 25% -45%. Combined chemotherapy including rituximab is recommended as a primary treatment.

In Korea, there are few studies on Waldenstrom's Macroglobulinemia, and a relatively large number of patients have studied the data of 71 patients in 2014, retrospectively. In the present study, we found that the combined chemotherapy regimen with rituximab significantly improved the overall response rates. Bortezomib may also be effective in the treatment of Waldenstrom's Macroglobulinemia. Based on this, clinical trials of combined chemotherapy with rituximab or dexamethasone have been conducted and 80-90% reported However, lenalidomide 15mg alone was administered, lenalidomide was effective in Waldenstrom's Macroglobulinemia with a 29% overall response rate.

The authors concluded that the combination therapy of rituximab, bortezomib, lenalidomide, and dexamethasone is an effective treatment regimen that can improve the overall response rate including complete remission. Patients with Waldenstrom's Macroglobulinemia diagnosed in Korea we planned this study to evaluate the efficacy and safety of lenalidomide maintenance therapy with chemotherapy with chemotherapy including rituximab, bortezomib, lenalidomide, and dexamethasone

ELIGIBILITY:
Inclusion Criteria:

1. Clinicopathological diagnosis of Waldenstrom's Macroglobulinemia
2. Patients who meet criteria for treatment using consensus panel criteria from the Second International Workshop on Waldenstrom's macroglobulinemia
3. Male or female patients aged ≥19 years
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
5. Patients must have measurable disease, IgM > 0.5g/dL
6. Appropriate bone marrow, liver, and kidney function
7. Patients who are able to understand oral and written instructions and who are able to comply with all requirements
8. Patients who provided agreement of subject consent (ICF) prior to initiation of clinical trial.
9. Female patients had to be post-menopausal for ≥1 year, surgically sterile, or practicing an effective method of birth control (as described in the protocol), and have a negative serum beta-human chorionic gonadotropin or urine pregnancy test at screening; they also had to agree to continue using birth control measures for ≥6 months after terminating treatment. Male patients had to agree to use an acceptable method of contraception for the duration of the study.

Exclusion Criteria:

1. Central nervous system involvement central nervous system (CNS) involvement by Waldenström's macroglobulinemia
2. Patients who have received rituximab, lenalidomide, or bortezomib
3. Patients who are allergic or hypersensitive to mouse (murine), chimeric, human or humanized proteins, lenalidomide, bortezomib
4. One of the following labs or more:

   * Absolute neutrophil count (ANC) <1,000 / μL
   * Platelet count <75,000 cells / μL when not transfused
   * Serum AST / ALT> 3 times the upper limit of normal
5. Renal failure requiring hemodialysis or peritoneal dialysis
6. Patients with uncontrolled severe heart disease
7. Patients who can not or do not want antithrombotic therapy
8. Patient has more than Grade 2 peripheral neuropathy on clinical examination during the screening period
9. Patient with a history of stroke or cerebral hemorrhage within 12 months bofore signing ICF
10. Patients who have been diagnosed with a currently unadjusted severe infection
11. Patients with known human immunodeficiency virus (HIV), hepatitis C infection
12. Patients diagnosed with malignancy within 5 years before signing ICF
13. Pregnant or lactating patients
14. Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor
15. Patients with acute diffuse invasive pulmonary disease and cardiovascular disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
survival | 2 years
  Response assessment in Waldenström macroglobulinaemia

CONTACTS AND LOCATIONS:
Overall Officials: HoSup Lee, Principal Investigator — KUGH
Locations (1):
- Kosin University Gospel Hospital, Busan, Sue-gu, South Korea

IPD SHARING:
Plan to Share IPD: No